CLINICAL TRIAL: NCT04889183
Title: SeMaglutide and Albuminuria Reduction Trial in Obese Individuals Without Diabetes
Acronym: SMART
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: University Medical Center Groningen (Other)
Collaborators: Novo Nordisk A/S (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 202100166; 2021-001247-27 (EudraCT Number)
Record Dates: First submitted 2021-05-06; First posted 2021-05-17 (Actual); Last update posted 2025-04-22 (Actual); Status verified 2024-11

CONDITIONS: Obesity; Albuminuria
Keywords: SMART; Semaglutide; UMCG; Lambers Heerspink
MeSH Terms: conditions — Obesity; Albuminuria | interventions — semaglutide

STUDY DESIGN:
Intervention Model Description: Randomized placebo controlled double-blind two arm parallel clinical trial
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Semaglutide (Experimental): Patients will be treated with semaglutide 3 mg/ml s.c. once weekly for 24 weeks. The starting dose of semaglutide will be 0.24 mg subcutaneous injection with increasing doses at 4, 8, 12, and 16 weeks to 0.5, 1,0, 1.7 and 2.4 mg once weekly.
  Interventions: Drug: Semaglutide
- Placebo (Placebo Comparator): Patients will receive a matching placebo s.c. once weekly.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Semaglutide — Patients will be treated for 24 weeks with semaglutide 3.0 mlg/ml s.c. once weekly. The starting dose of semaglutide will be 0.24 mg per week subcutaneous injection with increasing doses at 4, 8, 12, and 16 weeks to 0.5, 1,0, 1.7 and 2.4 mg.
  Arms: Semaglutide
Drug: Placebo — Patients will receive a matching placebo sc. once weekly during the treatment period of 24 weeks.
  Arms: Placebo

SUMMARY:
Study to assess the effects of weekly subcutaneous administration of the GLP1-RA semaglutide 2.4mg on kidney function parameters in obese/overweight individuals at high risk of CKD progression.

DETAILED DESCRIPTION:
Glucagon Like Peptide 1 Receptor Agonist (GLP1-RA) therapies have been introduced as antidiabetic drugs. In addition, GLP1-RA therapies reduce body weight, in patients with and without diabetes, without inducing hypoglycemia. Moreover, GLP1-RA reduce albuminuria in patients with type 2 diabetes, and liraglutide and semaglutide have been shown to improve various risk markers of CKD progression in non-diabetic obese individuals. It is therefore likely that these agents delay progression of kidney function decline in high risk obese/overweight, non-diabetic individuals.

The main objective of the study is to assess the albuminuria lowering effects of semaglutide 2.4 mg s.c. once weekly (Semaglutide 3 mg/ml) compared to placebo in obese/overweight non-diabetic individuals with elevated albuminuria. This will be tested in a 24-week randomized placebo controlled double-blind two arm parallel clinical trial with a 4 week wash-out period after 24 weeks double blind treatment to assess off drug effects.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years
* Body Mass index ≥ 27 kg/m2
* Albuminuria ≥ 30 mg/g and ≤ 3500 mg/g
* eGFR ≥ 25 ml/min/1.73m2
* Stable renal function prior to entry into the study defined as no more than 30% eGFR change in 3 months prior to enrolment
* Signed Informed Consent

Exclusion Criteria:

* Diagnosis with type 1 or type 2 Diabetes
* Hba1c ≥ 6.5% at screening
* Cardiovascular disease event in 3 months prior to enrollment
* Treatment with GLP-1 RA < 4 weeks prior to screening
* Uncontrolled thyroid disease TSH>6.0 mIU/L or <0.4 mIU/L at screening
* Acute pancreatitis < 180 days prior to screening
* History or presence of chronic pancreatitis
* Females of child-bearing potential who are pregnant, breast-feeding or have intention of becoming pregnant or are not using adequate contraceptive measures

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 125 (Actual)
Dates: Start 2022-03-14 (Actual); Primary Completion 2024-05-28 (Actual); Study Completion 2024-05-28 (Actual)

PRIMARY OUTCOMES:
Change from baseline to week 24 in urinary albumin:creatinine ratio (UACR) | Week 1 to week 24
  Measured in first morning void

SECONDARY OUTCOMES:
estimated glomerular filtration rate (eGFR) | Week 1 to week 24
  Change from baseline to week 24 in estimated glomerular filtration rate (eGFR)
Iohexol measured glomerular filtration rate (GFR) | Week 1 to week 24
  Change from baseline to week 24 in Iohexol measured glomerular filtration rate (GFR)
urinary albumin:creatinine ratio (UACR) during wash-out | week 24 to 28
  Change in urinary albumin:creatinine ratio (UACR) during wash-out
estimated glomerular filtration rate (eGFR) during wash-out | week 24 to 28
  Change in estimated glomerular filtration rate (eGFR) during wash-out
body weight | Week 1 to week 24
  Change from baseline to week 24 in body weight
hip circumference | Week 1 to week 24
  Change from baseline to week 24 in hip circumference
systolic and diastolic blood pressure | Week 1 to week 24
  Change from baseline to week 24 in systolic and diastolic blood pressure
extracellular fluid | Week 1 to week 24
  Change from baseline to week 24 in extracellular fluid as measured by bio-impedance
high sensitivity C-reactive protein (CRP) | Week 1 to week 24
  Change from baseline to week 24 in high sensitivity C-reactive protein (CRP)

CONTACTS AND LOCATIONS:
Locations (13):
- Canada (2):
  - University of Calgary, Calgary, Alberta
  - Division of Nephrology University Health Network, University of Toronto, Toronto, Ontario
- Germany (2):
  - University Hospital Erlangen, Erlangen
  - University Hospital Wuerzburg, Würzburg
- Netherlands (5):
  - Rijnstate, Arnhem, Gelderland
  - Isala, Zwolle, Overijssel
  - University Medical Center Groningen, Groningen, Provincie Groningen
  - Martini Ziekenhuis, Groningen, Provincie Groningen
  - Dept Internal Medicine, division of Nephrology Hospital Group Twente, Almelo
- Spain (4):
  - Vall d'Hebron University Hospital, Barcelona
  - Hospital Universitari de Bellvitge, Barcelona
  - Hospital Da Costa Burela, Lugo
  - Hospital Clínico Universitario, Valencia

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Apperloo EM, Gorriz JL, Soler MJ, Cigarran Guldris S, Cruzado JM, Puchades MJ, Lopez-Martinez M, Waanders F, Laverman GD, van der Aart-van der Beek A, Hoogenberg K, van Beek AP, Verhave J, Ahmed SB, Schmieder RE, Wanner C, Cherney DZI, Jongs N, Heerspink HJL. Semaglutide in patients with overweight or obesity and chronic kidney disease without diabetes: a randomized double-blind placebo-controlled clinical trial. Nat Med. 2025 Jan;31(1):278-285. doi: 10.1038/s41591-024-03327-6. Epub 2024 Oct 25. PMID 39455729